CLINICAL TRIAL: NCT05329350
Title: A Multicenter, International, Follow-up Study to Monitor the Efficacy and Safety of the Occlutech® Muscular Ventricular Septal Defect (mVSD) Occluder in Patients With Muscular Ventricular Septal Defects
Brief Title: Follow-up Study to Monitor the Efficacy and Safety of the Occlutech® mVSD Cases
Acronym: mVSD Registry
Status: Recruiting | Type: Observational
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2016_07
Record Dates: First submitted 2018-04-03; First posted 2022-04-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Muscular Ventricular Septal Defect
Keywords: mVSD Occluder; mVSD; Occlutech; Occlutech mVSD Occluder; Muscular ventricular septal defect closure; Transcatheter closure; Percutaneous occlusion; Periventricular closure; Post-market clinical follow-up; PMCF; Congenital heart defect; Structural heart disease intervention; Echocardiography follow-up
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- muscular ventricular septal defects: patients with muscular ventricular septal defects
  Interventions: Device: Occlutech muscular ventricular septal defect (mVSD) Occluder

INTERVENTIONS:
Device: Occlutech muscular ventricular septal defect (mVSD) Occluder — Percutaneous, transcatheter (catheter-based) non-surgical closure of a muscular ventricular septal defect (mVSD) using the Occlutech mVSD Occluder. The device is a self-expandable nitinol wire-mesh occluder with two retention discs connected by a flexible waist and incorporates polyester/PET patches to support defect occlusion and tissue ingrowth. Implantation is performed by experienced operators in a specialized cath lab according to the IFU and local routine; device sizing/selection is guided by imaging (e.g., transthoracic echocardiography, angiography, fluoroscopy). The system is deployed using compatible Occlutech delivery accessories (e.g., Occlutech Pistol Pusher and Occlutech Delivery Set [ODS v1 or ODS III], as applicable).

SUMMARY:
The Occlutech® mVSD is indicated for percutaneous occlusion of hemodynamically or clinically significant muscular ventricular septal defects.

The objectives of the study are:

* To confirm the efficacy of Occlutech mVSD in patients requiring transcatheter occlusion (closure) of muscular ventricular septal defects.
* To confirm the safety of Occlutech mVSD in patients requiring transcatheter occlusion (closure) of muscular ventricular septal defects.

DETAILED DESCRIPTION:
This is a multicenter, prospective, and retrospective, international, post-market clinical follow-up Study to monitor the efficacy and safety of the Occlutech mVSD in patients with muscular ventricular septal defects.

Safety and efficacy of implanted devices are assessed by echocardiography, vital signs, laboratory tests, and ECGs on Day 1 (within 48 hours post-procedure), follow-up 1 (between Day 30 and Day 60), follow-up 2 at 6 months (from Day 61 until 6 months), follow-up 3 at 1 year (from 6 months until 1 year), and follow-up 4 at 3 years (from 1 year until 3 years).

* Patients will be screened to determine eligibility for the registry based on inclusion/exclusion criteria, through their medical history, demographics, vital signs, clinical laboratory tests, performance of a 12 lead electrocardiogram (ECG) and echocardiography data.
* Participants are treated according to the instructions-for-use (IFU) of the device and according to clinical routine.
* Procedures are performed at sites having appropriate laboratory support and adequately trained imaging personnel. The procedure is performed by physicians with experience in a wide range of interventional cardiology and structural heart disease, including transcatheter patent ductus arteriosus, atrial septal defect, and ventricular septal defect (VSD) closures.

Recruitment will be open until 50 Patients have been enrolled. The primary safety endpoint is defined as the incidence of Serious Adverse Device Effects (SADEs) including procedure-related death, procedure-related stroke, ischemic stroke, systemic embolism, severe hemolysis, complete heart block requiring pacemaker implantation or device explanation, new onset of severe tricuspid regurgitation (TR), new the onset of severe aortic regurgitation (AR), severe right-left ventricular outflow obstruction (RVOTO-LVOTO), device embolization, cardiac tamponade, infective endocarditis, or vascular complications requiring open heart surgery up to 1 year after the mVSD closure procedure.

The primary efficacy endpoints will include data obtained 1 year after the mVSD closure procedure for successful implantation of the device with a proper closure of the mVSD (defined as the reduction in muscular ventricular septal shunt to trivial or no shunt at all, as assessed by echocardiography pre- vs post-implantation).

ELIGIBILITY:
Inclusion Criteria

* A participant will be eligible for study participation if he/she meets the indication and area of application as laid down in the IFU. The Occlutech mVSD is indicated for percutaneous occlusion of hemodynamically or clinically significant muscular ventricular septal defects.
* Any age
* Male or female.
* Patients understand the nature of the study and provide their informed consent to participation.
* Patients willing and able to attend the follow-up visits and procedures foreseen by study CIP.

Contraindication

* Hemodynamically relevant VSD shunt
* Congestive heart insufficiency
* Recurrent respiratory infections
* Failure to thrive.
* Significant left ventricle (LV) enlargement
* Significant left atrium (LA) enlargement
* Other clinical indication

Exclusion Criteria

The device is contraindicated for participants known to have any of the following:

⦁Active bacterial infections

* Active infection at the time of implantation
* Allergy to antiplatelet or anticoagulant therapy
* Allergy to nickel and/or titanium and/or nickel/titanium-based materials
* Any type of serious infection 1 month before the procedure
* The aortic rim of less than 2 mm
* Demonstrated intracardiac thrombi on echocardiography
* Malignancy where life expectancy is less than 3 years
* mVSD diameter > 20 mm
* Perimembranous VSD

Post-MI VSD

* Recent myocardial infarction or a surgical bypass operation in the last 30 days
* Sepsis (local or generalized)
* Septal thickness > 7 mm in the area of the Occluder placement

Ages: 3 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients of any age with a hemodynamically or clinically significant muscular ventricular septal defect (mVSD) who are candidates for non-surgical closure with the Occlutech mVSD Occluder in routine clinical practice (predominantly pediatric patients). Eligibility is confirmed based on protocol-defined inclusion/exclusion criteria and baseline clinical assessment, including medical history, demographics, vital signs, ECG and echocardiography; laboratory tests may be performed according to local standard of care.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint | 1 year
  The primary safety endpoint is defined as the incidence of Serious Adverse Device Effects (SADEs) including procedure-related death, procedure-related stroke, ischemic stroke, systemic embolism, severe hemolysis, complete heart block requiring pacemaker implantation or device explanation, new onset of severe tricuspid regurgitation (TR), new the onset of severe aortic regurgitation (AR), severe right-left ventricular outflow obstruction (RVOTO-LVOTO), device embolization, cardiac tamponade, infective endocarditis, or vascular complications requiring open heart surgery up to 1 year after the mVSD closure procedure.
The primary efficacy endpoint | 1 year
  The primary efficacy endpoints will include data obtained 1 year after the mVSD closure procedure for successful implantation of the device with a proper closure of the mVSD (defined as the reduction in muscular ventricular septal shunt to trivial or no shunt at all, as assessed by echocardiography pre- vs post-implantation).

CONTACTS AND LOCATIONS:
Locations (5):
- Children's Health Ireland, Dublin, Ireland
- Turkey (Türkiye) (4):
  - İzmir Şehir Hastanesi, Izmir, Bayraklı
  - Eskişehir Osmangazi Üniversite Hastanesi, Eskişehir, Odunpazarı
  - Dicle Üniversitesi Tıp Fakültesi Hastanesi, Diyarbakır, Sur
  - Gaziantep Unıversıty Hospital, Gaziantep, Şehitkamil

IPD SHARING:
Plan to Share IPD: Undecided